CLINICAL TRIAL: NCT07290335
Title: Optimizing Strategies to Maximize Patient Recruitment Yield
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other); Georgia Clinical and Translational Science Alliance (GaCTSA) (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Neal Dickert, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P013508; UL1TR002378 (NIH)
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Recruitment
Keywords: Research recruitment; Patient portal-based communication
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline (control) message (Active Comparator): Patients in the Emory Healthcare system, who have not opted out of research contact, receiving MyChart messaging for research recruitment using the current standard template.
  Interventions: Behavioral: Baseline (control) message
- Positively-valenced message (Experimental): Patients in the Emory Healthcare system, who have not opted out of research contact, receiving MyChart messaging for research recruitment using a template with inclusion of positively-valenced language describing the study's value.
  Interventions: Behavioral: Positively-valenced message
- Payment-inclusive message (Experimental): Patients in the Emory Healthcare system, who have not opted out of research contact, receiving MyChart messaging for research recruitment using a template containing information about payment to participants.
  Interventions: Behavioral: Payment-inclusive message
- Positively-valenced, payment-inclusive message (Experimental): Patients in the Emory Healthcare system, who have not opted out of research contact, receiving MyChart messaging for research recruitment using a template with both positively-valenced language and payment information.
  Interventions: Behavioral: Positively-valenced, payment-inclusive message

INTERVENTIONS:
Behavioral: Baseline (control) message — The MyChart study recruitment program will send a message based on the current template, which is a brief message with a neutral tone.
  Arms: Baseline (control) message
Behavioral: Positively-valenced message — The MyChart study recruitment program will send a message based on a template that contains positively-valenced language related to the value/importance of the study.
  Arms: Positively-valenced message
Behavioral: Payment-inclusive message — The MyChart study recruitment program will send a message based on a template that includes more detailed information about participant payment.
  Arms: Payment-inclusive message
Behavioral: Positively-valenced, payment-inclusive message — The MyChart study recruitment program will send a message based on a template that includes both positively-valenced language and detailed information about participant payment.
  Arms: Positively-valenced, payment-inclusive message

SUMMARY:
This platform trial aims to evaluate the effectiveness of different messaging strategies within a MyChart messaging program for research recruitment. MyChart is a patient portal system within the Electronic Medical Record (EMR), and messages can be sent directly to patients about research opportunities.

DETAILED DESCRIPTION:
Recruitment of participants presents a significant and persistent bottle neck in the research process. Failure to reach participant enrollment targets may delay or halt study progression, wasting limited resources. Insufficient rates of participant accrual are the leading cause for termination among clinical trials with results posted on ClinicalTrials.gov. Additionally, studies must enroll representative samples to ensure generalizability and comply with NIH guidelines. Investigators often cite recruitment difficulties - including lack of interest, difficulty reaching specific populations, and limited resources - to explain failure to reach enrollment goals. However, these recruitment difficulties may not actually be due to a lack of willingness to participate among eligible patients. A national survey conducted by Harris Interactive in 2001 found that 85% of patients were either unaware or unsure that participation in a clinical trial was an option at the time of diagnosis. 75% of these patients said they would have been willing to enroll had they known it was possible. Innovation in recruitment is sorely needed to make recruitment more efficient and more representative.

In recent years, researchers have begun to leverage patient portals and electronic health records (EHRs) for recruitment. This method allows for engagement of broad populations within a health system in a cost-effective way. Emerging evidence of EHR recruitment shows promise. The researchers of this study have examined the use of EHR recruitment to identify and contact eligible patients via MyChart direct-to-patient messaging across a range studies within Emory Healthcare. Having completed a pilot program within the Emory system, this service is now available to all Emory investigators for whom MyChart recruitment is appropriate.

While the feasibility of MyChart messaging has been documented, little is known about best practices for how recruitment messages should be designed. There are, however, good reasons to believe that how messages are designed and framed may impact potential participants' responses to them.

This project is a platform trial that will allow for serial testing of various aspects of portal-based messaging. Consistent with platform trial design, the researchers will use a common set of outcome measures across various studies, and the portal-based messaging strategy allows for easy randomization (generally at the patient level) of patients to specific messaging approaches.

In the context of broader use of MyChart messaging, the researchers have designed this study to examine the impact of message design on patients' responses. Specifically, this study will examine the impact of including positively-valenced language that describes the value of the study and the impact of inclusion of information regarding any payments that participants will receive in the study. Both of these factors are ones that are grounded in behavioral economics and may be meaningful to potential participants.

The first proposed trial will involve randomly assigning patients who are identified as potentially eligible for studies using the MyChart recruitment mechanism to receive a recruitment message using 1 of 4 templates: 1) the current standard template; 2) a template with inclusion of positively-valenced language describing the study's value; 3) a template containing information about payment to participants; and 4) a template with both positively-valenced language and payment information. For all studies using the MyChart mechanism, all 4 messages will be created, and assignment will be done based on the last two digits of the patient's medical record number (MRN).

The primary endpoint is the rate at which individuals respond that they are interested in participating in the study to which they are invited. Additionally, this study will examine the non-response rate and the rate of individuals responding that they are not interested in the study. It will also track the rate at which individuals exposed to a MyChart recruitment message change their permission settings for contact about research opportunities. Study teams whose study invitations are used in this trial will be contacted about the rate of enrollment among patients who responded as "interested" to the message so that the researchers can estimate enrollment rate within each intervention group. Finally, select patients will participate in short interviews to understand their impressions of the message they were sent and their attitudes towards research more generally.

ELIGIBILITY:
Inclusion Criteria for primary studies that are recruiting participants:

* All studies using the MyChart recruitment service are eligible, including both clinical trials and observational studies.

Exclusion Criterion for primary studies that are recruiting participants:

* Not using MyChart for recruitment.
* At least 500 messages sent, 125 for each arm

Inclusion Criteria for patients:

* All patients receiving messages via MyChart will be included
* Potential eligibility for a study using MyChart requirement based on the planned query/criteria for that study.

Exclusion Criteria for patients:

* Minor
* Excluded from primary study that is recruiting participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of "interested" response to recruitment messages | Month 12
  The primary endpoint is the rate at which individuals respond that they are interested in participating in the study to which they are invited. The primary outcome is a binary variable of "interested" response.

SECONDARY OUTCOMES:
Rate of non-response | Month 12
  This study will examine the rate of non-response to recruitment messages.
Rate of "not interested" responses | Month 12
  This study will examine the rate of individuals responding that they are not interested in the study.
Rate of change in MyChart permissions to contact | Month 12
  This study will examine the rate at which individuals exposed to a MyChart recruitment message change their permission settings for contact about research opportunities.
Rate of enrollment among "interested" patients | Month 12
  Study teams whose study invitations are used in this trial will be contacted about the rate of enrollment among patients who responded as "interested" to the message.
Patient impressions on recruitment messages | Month 12
  Some patients will participate in short interviews to understand their impressions of the message they were sent. Qualitative data are collected during the interviews and there is not a standardized questionnaire or scale that will be used.
Patient impressions on research in general | Month 12
  Some patients will participate in short interviews to understand their attitudes towards research more generally. Qualitative data are collected during the interviews and there is not a standardized questionnaire or scale that will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Dickert, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Healthcare System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available for sharing. This will include deidentified participant-level demographic characteristics, intervention assignment, and enrollment/non-enrollment status within the parent trial. This will include a de-identified data spreadsheet, readme file, and a data dictionary.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be uploaded into a repository at the time of publication of findings from this study.
Access Criteria: Deidentified participant-level data and associated metadata will be uploaded into the Emory Dataverse (https://dataverse.unc.edu/dataverse/Emory).